CLINICAL TRIAL: NCT05307783
Title: A Multicenter Observational Study to Evaluate Outcomes of EmboCube Gelatin Embolization to Control Bleeding or Hemorrhaging
Brief Title: EmboCube Gelatin Embolization to Control Bleeding or Hemorrhaging
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EGE-P4-21-01
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhage; Bleeding Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: EmboCube Embolization Gelatin — EmboCube is a uniformly cut gelatin foam pre-loaded into a syringe, indicated for use in embolization of blood vessels to occlude blood flow to control bleeding/hemorrhaging in the peripheral vasculature

SUMMARY:
This is a multicenter, observational study of the use of EmboCube Embolization Gelatin to control hemorrhaging and bleeding. The study is designed to enable the collection, analysis, and reporting of data from "real-world" use of EmboCube used in accordance with the Instructions for Use (IFU) associated with the product's CE Mark approval.

Data collection will include that relating to safety and effectiveness and the period of observation during which data will be collected will extend from the index procedure through 28 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subject requires embolization and is suitable for treatment with EmboCube in accordance with device Instructions For Use for the treatment of bleeding or hemorrhage.
3. Subject provides written informed consent to study data collection.

Exclusion Criteria:

1. Bleeding site in the neck, head, or brain.
2. Subject has co-morbidity with survival prognosis of less than 30 days, in the opinion of the treating physician
3. In the investigator's opinion, participation in the study may not be in the subject's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are treated with EmboCube to control bleeding or hemorrhage in accordance with the current approved CE Mark indication for use (IFU) as stated in the IFU.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - South Western Sydney Local Health District, Liverpool
  - Alfred Health, Sydney
- France (2):
  - Centre Hospitalier Universitaire de Nîmes - Caremeau, Nîmes
  - HEGP, Paris

REFERENCES:
- [Derived] Pellerin O, Frandon J, Schlaphoff G, Copping R, Dean C, Clements W. A multicenter prospective study evaluating use of EmboCube Embolization Gelatin alone or in combination with other embolic agents to control bleeding. CVIR Endovasc. 2025 May 31;8(1):50. doi: 10.1186/s42155-025-00571-w. PMID 40448890

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: Treated with EmboCube Embolization Gelatin
Period: Overall Study
Arm/Group | Device
Started | 101
Completed | 90
Not Completed | 11
Not completed — Death | 7
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Device
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (20.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American / Black | 2
  Race: Asian | 6
  Race: Caucasian/ White | 40
  Race: Pacific Islander | 5
  Race: Other | 23
  Race: Not reported / Refuse to disclose | 25
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 50
  France | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success: Cessation of Bleeding up to 24 Hours
Description: The primary performance endpoint will be clinical success defined as cessation of bleeding post-embolization and absence of rebleeding at the treated site requiring reintervention (repeat embolization or additional surgery), within 24 hours.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 100

2. Primary Outcome: Number of Participants Without Device and Procedure-related AEs (Incidence of Device and Procedure-related AEs)
Description: Absence of unanticipated serious adverse device effects within 24 hours.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 101

ADVERSE EVENTS:
Time Frame: Data collection included endpoints relating to safety and effectiveness during the period from index procedure through 28 days post-procedure.
Arm/Group | Device
All-Cause Mortality (participants affected / at risk) | 7/101
Serious Adverse Events (participants affected / at risk) | 12/101
Other Adverse Events (participants affected / at risk) | 3/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=101)
Bleeding complication (Vascular disorders) | 1 (1)
Hematoma (Surgical and medical procedures) | 1 (1)
Hemorrhage (Vascular disorders) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Hematoma of the left kidney (Vascular disorders) | 1 (1)
Progressive deterioration of liver function (Hepatobiliary disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Cirrhosis (Hepatobiliary disorders) | 1 (1)
Ischemic colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=101)
Aneurysm (Vascular disorders) | 1 (1)
Renal failure/renal insufficiency (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT05307783/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT05307783/SAP_001.pdf